CLINICAL TRIAL: NCT04854707
Title: An Observational Study "FOLLITROPIN" Comparing the Efficacy of Follitropin Alpha Biosimilar: the Real-world Data
Brief Title: An Observational Study of Follitropin Alpha Biosimilar: the Real-world Data
Status: Completed | Type: Observational
Sponsor: IVFarma LLC (Industry)
Collaborators: Institute for Preventive and Social Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: IVF-2020
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Reproductive Issues; Reproductive Disorder; Fertility Disorders; Fertility Issues; Gynecologic Disease; IVF
Keywords: follitropin alpha; follicle-stimulating hormone; in vitro fertilization; assisted reproductive technologies; biosimilar; follitropin alfa; real-world data
MeSH Terms: conditions — Infertility; Genital Diseases, Female | interventions — follitropin alfa; Biosimilar Pharmaceuticals; Menotropins; follitropin beta; Luteinizing Hormone, beta Subunit; follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH: The ovarian stimulation (OS) protocols included monotherapy protocols with using follitropin alpha biosimilar only and antagonists/agonists of of gonadotropin-releasing hormone (GnRH): ganirelix, cetrorelix, triptorelin, buserelin.
  Interventions: Drug: Follitropin Alfa
- Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH: The OS protocols included: mixed protocols (recombinant with addition of urinary-derived gonadotropins) and antagonists/agonists of GnRH (ganirelix, cetrorelix, triptorelin, buserelin), where follitropin alpha biosimilar used for at least 5 days during OS.
  Interventions: Drug: Follicle Stimulating Hormone/Luteinizing Hormone
- Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH: The OS protocols included: monotherapy protocols with using only follitropin alpha biosimilar and antagonists of GnRH.
  Interventions: Drug: Follitropin Alfa
- Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH: The OS protocol included: monotherapy protocols with using only follitropin alpha biosimilar and agonists of GnRH.
  Interventions: Drug: Follitropin Alfa
- The overall protocols: The OS protocols included: (1) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH, (2) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH
  Interventions: Drug: Follicle Stimulating Hormone/Luteinizing Hormone

INTERVENTIONS:
Drug: Follitropin Alfa — Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using antagonists of GnRH or agonist of GnRH.
  Other Names: Primapur; Biosimilar
  Groups: Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH
Drug: Follicle Stimulating Hormone/Luteinizing Hormone — Subcutaneous injection of follitropin alpha biosimilar, with daily dose 100-300 IU for at least 5 days, than added another gonadotropin for a maximum of 10 days, using antagonists of GnRH or agonist of GnRH.
  Other Names: Follitropin beta; Follitropin alfa + Lutropin alfa; Corifollitropin alfa; Menotropins; Follitropin alfa; Follitropin alfa biosimilar
  Groups: Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH
Drug: Follitropin Alfa — Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using antagonists of GnRH only for suppression.
  Other Names: Primapur; Biosimilar; Follitropin alfa biosimilar
  Groups: Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH
Drug: Follitropin Alfa — Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using agonists of GnRH only for suppression.
  Other Names: Primapur; Biosimilar; Follitropin alfa biosimilar
  Groups: Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH
Drug: Follicle Stimulating Hormone/Luteinizing Hormone — Overall ovarian stimulation protocols with follitropin alpha biosimilar for at least 5 days+other recombinant and menotropins and short (antagonists of GnRH) or long protocol (agonist of GnRH).
  Other Names: Follitropin beta; Corifollitropin alfa; Follitropin alfa + Lutropin alfa; Menotropins; Follitropin alfa biosimilar; Follitropin alfa
  Groups: The overall protocols

SUMMARY:
Aim to investigate the efficacy of follitropin alpha biosimilar therapy (Primapur®) in nonselected real-world population.

DETAILED DESCRIPTION:
A retrospective observational anonymized cohort study of follitropin alpha biosimilar (Primapur®) as a pre-filled pen injector with a dose adjustment of 5 IU, aimed to investigate its efficacy and safety in a nonselected population with indications to assisted reproductive technologies (ART) was carried out. The ovarian stimulation (OS) protocols included:

monotherapy protocols with using only Primapur®; mixed protocols (recombinant and urinary-derived gonadotropins); short protocols with using antagonists of gonadotropin-releasing hormone (GnRH) and long protocols with GnRH agonists. The stimulation protocols were analyzed with Primapur® application for at least 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Women with established causes of infertility and indications for the use of ART methods, according to the Order of the Ministry of Health of the Russian Federation "On the use of assisted reproductive technologies, contraindications and limitations to their use" No. 107 n dated August 30, 2012.
* Infertility due to female and/or male factor.
* Presence of ovaries accessible for aspiration of follicles.
* Anatomical and functional capability of uterus to bear pregnancy.

Exclusion Criteria:

* Women with established contraindications to the use of ART methods, according to the Order of the Ministry of Health of the Russian Federation "On the use of assisted reproductive technologies, contraindications and limitations to their use" No. 107 n dated August 30, 2012.
* Presence of pregnancy
* Hypersensitivity to follitropin alfa or excipients.
* Ovarian cysts (not associated with polycystic ovarian syndrome), uterine hemorrhage of unclear etiology
* Premature ovarian failure
* Presence of clinically significant systemic disease
* Presence of chronic cardiovascular, hepatic, renal or pulmonary disease
* Neoplasia
* Narcomania, alcoholism

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women aged 20-43 with established causes of infertility and indications for the use of assisted reproductive technologies (ART) and ovarian stimulation with follitropin alpha.
Sampling Method: Non-Probability Sample
Enrollment: 5484 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilorom Kamilova, PhD, Principal Investigator — MD Medical Group
Locations (35):
- Russia (35):
  - Center for reproductive medicine, Barnaul, Barnaul
  - Center for reproductive medicine, Irkutsk, Irkutsk
  - Clinic "Mother and Child" Kazan, Kazan'
  - Clinic "Mother and Child" Kostroma, Kostroma
  - Clinic "Mother and Child" Krasnodar, Krasnodar
  - Center for reproductive medicine, Krasnoyarsk, Krasnoyarsk
  - AltraVita IVF clinic, Moscow
  - Center of Reproductive Medicine and Genetics "Nova Clinic", Moscow
  - Clinic "Mather and Child" Lefortovo, Moscow
  - Clinic "Mather and Child" Savelovskaya, Moscow
  - Clinic "Mother and Child" Khodynskoe Pole, Moscow
  - Clinic "Mother and Child" Kuntsevo, Moscow
  - Clinic "Mother and Child" South-West, Moscow
  - Clinical Hospital MD GROUP (Perinatal Center on Sevastopolskiy), Moscow
  - Clinical Hospital Lapino, Moscow Oblast
  - Clinic "Mother and Child", Nizhny Novgorod
  - Medika-2, Novokuznetsk
  - Center for reproductive medicine, Novosibirsk, Novosibirsk
  - Clinical Hospital "Avicenna", Novosibirsk
  - Ceter for reproductive medicine, Omsk, Omsk
  - Clinic "Mother and Child" Perm, Perm
  - Clinic "Mother and Child" Rostov-on-Don, Rostov-on-Don
  - Clinic "Mather and Child", Ryazan
  - "Genesis" Reproduction Centre, Saint Petersburg
  - Clinic "Mother and Child" Saint-Petersburg, Saint Petersburg
  - Clinical Hospital "Mother and Child", Samara
  - Clinic "Mather and Child" Tula, Tula
  - Clinical Hospital "Mother and Child", Tyumen
  - Clinical Hospital "Mother and Child", Ufa
  - Clinic "Mother and Child" Vladimir, Vladimir
  - Clinic "Mather and Child" Vladivostok, Vladivostok
  - Clinic "Mother and Child" Volgograd, Volgograd
  - Clinic "Mother and Child" Voronezh, Voronezh
  - Clinic "Mother and Child" Yaroslavl, Yaroslavl
  - Clinical Institute of Reproductive Medicine, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] M Polzikov, D Kamilova, M Ovchinnikova, E Mayasina, K Boyarsky, S Nikitin, I Bendusov, M Ganikhina, Z Barakhoeva, E Osina, E Ablyaeva, D Khetagurova, T Ushakova, D Blinov, P-669 "Follitropin": A retrospective, observational study comparing the efficacy of follitropin alpha biosimilar therapy in different ovarian stimulation protocols: real-world data, Human Reproduction, Volume 36, Issue Supplement_1, July 2021, deab130.668. https://doi.org/10.1093/humrep/deab130.668
- [Result] Kamilova D.P., Ovchinnikova M.M., Ablyaeva E.S., Leviashvili M.M., Stuleva N.S., Broitman E.V., Ganikhina M.A., Mayasina E.N., Iskhakova L.F., Boyarskiy K.Yu., Ovsyannikova E.N., Barakhoeva Z.B., Nikitin S.V., Bendusov I.A., Fetisova Yu.A., Yudina M.A., Tararashkina E.S., Khetagurova D.T., Blinov D.V., Polzikov M.A. An observational study "FOLLITROPIN" comparing the efficacy of follitropin alpha biosimilar: the real-world data. Obstetrics, Gynecology and Reproduction. 2021;15(1):5-21. (In Russ.) https://doi.org/10.17749/2313-7347/ob.gyn.rep.2021.212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All of the analysed subjects underwent OS using GnRH antagonist/agonist protocols, with no restrictions on the OS protocol or food supplements/vitamins.
Period: Overall Study
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH
Started | 2625 | 2183 | 676
Completed | 2547 | 2124 | 646
Not Completed | 78 | 59 | 30
Not completed — Lack of Efficacy | 78 | 59 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | Total
Number analyzed (Participants) | 2625 | 2183 | 676 | 5484
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (4.8) | 32.9 (4.6) | 33.1 (4.9) | 33.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2625 | 2183 | 676 | 5484
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2625 | 2183 | 676 | 5484
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 2625 | 2183 | 676 | 5484
Body Mass Index (BMI), kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (4.7) | 23.7 (4.6) | 23.1 (4.5) | 23.8 (5.7)
Duration of infertility, years [Mean (Standard Deviation); unit: years] | 5.7 (4.1) | 5.4 (4.3) | 5.6 (3.8) | 5.6 (4.2)
IVF attempt [Mean (Standard Deviation); unit: number of IVF attempts] | 1.4 (0.7) | 1.2 (0.5) | 1.4 (0.9) | 1.3 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: The total number of retrieved oocytes at the day of ovum pick-up. No more than 37 hours from the introduction of the ovulation inducer (HCG or GnRH-agonist).
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) the analysed population was: (1) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH - 2625 participants (lack of efficacy: 78 participants, the analysed population was 2547 participants); (2) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH - 2859 participants (lack of efficacy: 89, the analysed population was 2770); (3) Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH - 2183 participants (lack of efficacy: 59, the analysed population was 2124) and (4) Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH - 676 participants (lack of efficacy: 30, the analysed population was 646).
Time Frame: From date of start of ovarian stimulation with follitropin alpha up to 15 days
Population: Arm "Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH" is combined group for primary and secondary outcome measures and consist of patients from "Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH" and "Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH".
Measure: Mean (Standard Deviation); unit: The total number of retrieved oocytes
Groups:
- Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH: The OS protocols included: mixed protocols (recombinant with addition of urinary-derived gonadotropins) and antagonists/agonists of GnRH (ganirelix, cetrorelix, triptorelin, buserelin), where follitropin alpha biosimilar used for at least 5 days during OS.
  Follicle Stimulating Hormone/Luteinizing Hormone: Subcutaneous injection of follitropin alpha biosimilar, with daily dose 100-300 IU for at least 5 days, than added another gonadotropin for a maximum of 10 days, using antagonists of GnRH or agonist of GnRH.
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) in 78 participants (or 3%), the analysed population was 2547 participants.
- Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH: The ovarian stimulation (OS) protocols included monotherapy protocols with using follitropin alpha biosimilar only and antagonists/agonists of of gonadotropin-releasing hormone (GnRH): ganirelix, cetrorelix, triptorelin, buserelin.
  Follitropin Alfa: Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using antagonists of GnRH or agonist of GnRH.
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) in 89 participants (or 3,1%), the analysed population was 2770 participants.
- Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH: The OS protocols included: monotherapy protocols with using only follitropin alpha biosimilar and antagonists of GnRH.
  Follitropin Alfa: Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using antagonists of GnRH only for suppression.
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) in 59 participants (or 2,7%), the analysed population was 2124 participants.
- Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH: The OS protocol included: monotherapy protocols with using only follitropin alpha biosimilar and agonists of GnRH.
  Follitropin Alfa: Subcutaneous injection of follitropin alpha biosimilar only, with daily dose 100-300 IU for 10 days, maximum of 15 days, using agonists of GnRH only for suppression.
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) in 30 participants (or 4,4%), the analysed population was 646 participants.
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | The Overall Protocols
Number analyzed (Participants) | 2547 | 2770 | 2124 | 646 | 5317
The total number of retrieved oocytes | 8.6 (6.8) | 10.3 (7.4) | 10.5 (7.5) | 9.6 (7.0) | 9.5 (7.2)
Statistical Analysis 1: Comparison: Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH; Test type: Other; p = 0.032, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Percentage of Participants With Ongoing Clinical Pregnancy Per Embryo Transfer
Description: Ongoing clinical pregnancy per embryo transfer (detection of gestational sac and heartbeat from 6 weeks after transfer), n (ongoing pregnancy rate per transfer with known outcome, %).
  Due to delayed embryo transfers, the analysed population for "Ongoing clinical pregnancy per embryo transfer" was: (1) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH - 2007 embryo transfers (1542 with known outcome); (2) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH - 2213 embryo transfers (1800 with known outcome); (3) Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH - 1809 embryo transfers (1466 with known outcome) and (4) Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH - 404 embryo transfers (334 with known outcome).
Time Frame: At least 6 weeks after embryo transfer
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percetnage of patients (%)
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | The Overall Protocols
Number analyzed (Participants) | 1542 | 1800 | 1466 | 334 | 3342
Percetnage of patients (%) | 39.3 [36.9 to 41.7] | 37.6 [35.3 to 39.8] | 37.9 [35.5 to 40.5] | 35.9 [30.8 to 41.1] | 38.4 [35.9 to 40.2]
Statistical Analysis 1: Comparison: Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH; 95% Confidence intervals (CIs) of point estimates were calculated using the exact binominal distribution (Clopper-Pearson method) for proportions; Test type: Other; p = 0.314, Chi-squared; z-value = 1; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.0161 to 0.0501]
Statistical Analysis 2: Comparison: Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.482, Chi-squared; Mean Difference (Final Values) = 0.0207, 95% CI 2-sided [-0.0369 to 0.0782]

3. Secondary Outcome: Number of Mature Oocytes
Description: Mature oocytes (MII stage of development).
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) the analysed population was: (1) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH - 2625 participants (lack of efficacy: 78 participants, the analysed population was 2547 participants); (2) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH - 2859 participants (lack of efficacy: 89, the analysed population was 2770); (3) Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH - 2183 participants (lack of efficacy: 59, the analysed population was 2124) and (4) Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH - 676 participants (lack of efficacy: 30, the analysed population was 646).
Time Frame: From date of start of ovarian stimulation with follitropin alpha up to 15 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of mature oocytes
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | The Overall Protocols
Number analyzed (Participants) | 2547 | 2770 | 2124 | 646 | 5317
Number of mature oocytes | 6.7 (6.2) | 7.7 (6.9) | 7.6 (6.9) | 6.7 (5.7) | 6.8 (6.6)
Statistical Analysis 1: Comparison: Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Fertilized Oocytes
Description: Fertilization rate (FR) is percentage of transformation of oocytes into two pronuclei (presence of two pronuclei: zygotes with 2PN).
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) the analysed population was: (1) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH - 2625 participants (lack of efficacy: 78 participants, the analysed population was 2547 participants); (2) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH - 2859 participants (lack of efficacy: 89, the analysed population was 2770); (3) Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH - 2183 participants (lack of efficacy: 59, the analysed population was 2124) and (4) Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH - 676 participants (lack of efficacy: 30, the analysed population was 646).
Time Frame: From date of start of ovarian stimulation with follitropin alpha up to 16 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: zygotes with 2PN
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | The Overall Protocols
Number analyzed (Participants) | 2547 | 2770 | 2124 | 646 | 5317
zygotes with 2PN | 5.8 (5.2) | 7.2 (6.2) | 7.3 (6.3) | 5.7 (5.0) | 6.1 (5.8)
Statistical Analysis 1: Comparison: Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Total Dose of Follitropin Alpha Biosimilar Protocol, IU
Description: Mean dose of follitropin alpha biosimilar for ovarian stimulation.
  Due to lack of efficacy of the therapy (ovarian stimulation was not completed and oocytes were not retrieved) the analysed population was: (1) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH - 2625 participants (lack of efficacy: 78 participants, the analysed population was 2547 participants); (2) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH - 2859 participants (lack of efficacy: 89, the analysed population was 2770); (3) Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH - 2183 participants (lack of efficacy: 59, the analysed population was 2124) and (4) Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH - 676 participants (lack of efficacy: 30, the analysed population was 646).
Time Frame: From date of start of ovarian stimulation with follitropin alpha up to 16 days
Measure: Mean (Standard Deviation); unit: IU (International Units)
Arm/Group | Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH | Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH | The Overall Protocols
Number analyzed (Participants) | 2547 | 2770 | 2124 | 646 | 5317
IU (International Units) | 1672 (568) | 1919 (639) | 1952 (621) | 1711 (680) | 1825 (647)
Statistical Analysis 1: Comparison: Mixed Protocols: Recombinant and Urinary-derived Gonadotropins and Antagonists/Agonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists/Agonists of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Monoprotocols: Follitropin Alpha Biosimilar Only and Antagonists of GnRH vs Monoprotocols: Follitropin Alpha Biosimilar Only and Agonist of GnRH; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The time frame was 20 days: ovarian stimulation (up to 15 days) till the day of embryo transfer (up to 5 days).
Description: Serious adverse events collection (hospitalizations). Due to overall ovarian stimulation protocols consist of follitropin alpha biosimilar treatment for at least 5 days, the adverse events were combined in one group ("Overall protocols"). The questionary was not include the enquiry for exact description of ovarian stimulation protocol (or treatment).
Groups:
- The Overall Protocols: The overall protocols (groups) were combined and analysed for Serious Adverse Events and other (not including serious) adverse events.
  Due to overall ovarian stimulation protocols consist of follitropin alpha biosimilar treatment for at least 5 days, the adverse events were combined in one group to analyse the safety of follitropin alpha biosimilar treatment not in relation to protocol of ovarian stimulation and other medication.
Arm/Group | The Overall Protocols
All-Cause Mortality (participants affected / at risk) | 0/5484
Serious Adverse Events (participants affected / at risk) | 0/5484
Other Adverse Events (participants affected / at risk) | 657/5484
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Overall Protocols (N=5484)
Injection site pain (Skin and subcutaneous tissue disorders) | 657 (657) — Injection site pain was classified as skin and subcutaneous tissue disorders and included redness, pain, bruising and irritation without differentiation.

LIMITATIONS AND CAVEATS:
The real-world patient data analysed in this study were representative, showing the ability of follitropin biosimilars to develop both folliculogenesis and clinical pregnancy in a nonselected population. Additional comparative studies are needed to confirm the efficacy of the biosimilars in patients with classified types of infertility causes, including unexplained infertility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04854707/Prot_SAP_000.pdf